CLINICAL TRIAL: NCT00772694
Title: Sorafenib (NEXAVAR) Monotherapy in Patients With Inoperable/Recurrent Germ Cell Carcinoma Refractory to Chemotherapy
Brief Title: Sorafenib Monotherapy in Inoperable/Recurrent Germ Cell Carcinoma Refractory to Chemotherapy
Acronym: GCT
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fondation Wygrajmy Zdrowie (Other)
Responsible Party: dr Iwona Skoneczna, Fondation Wygrajmy Zdrowie
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 12602; PL/ 183/UR/CEBK/04/08; EudraCT 2007-007599-40
Record Dates: First submitted 2008-10-14; First posted 2008-10-15 (Estimated); Last update posted 2008-10-24 (Estimated); Status verified 2008-10

CONDITIONS: Testicular Cancer
Keywords: testicular cancer; germ cell cancer; sorafenib
MeSH Terms: conditions — Testicular Neoplasms; Neoplasms, Germ Cell and Embryonal | interventions — Sorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- sorafenib (Experimental): drug
  Interventions: Drug: sorafenib

INTERVENTIONS:
Drug: sorafenib — tablets 200mg, 400mg bid continuously in 4-week cycles
  Other Names: Nexavar

SUMMARY:
Germ cell tumors, a relatively rare disease, but most common malignancy in young males, occur most frequently in testis. The incidence is about 1%, but is increasing in the majority of developed countries. The testicular cancer is an extremely important oncological condition due to his high rate of 80-90% of curability, which can be achieved by combination of chemotherapy and surgery.

Some of 20-30% of patients will experience disease progression after first line cisplatin-based chemotherapy and salvage 2nd line conventional-dose cisplatin-based salvage chemotherapy will result in long term remissions in < 50% of patients (VeIP - vinblastine, ifosfamide, cisplatin, VIP/PEI - ifosfamide, etoposide, cisplatin, TIP - paclitaxel, ifosfamide, cisplatin). In multiple relapsed patients the 3rd line chemotherapy can induce remission in up to 40% (gemcitabine, oxaliplatin), 23% RR (TG - paclitaxel, gemcitabine), 20% CR (IPO - irinotecan, paclitaxel, oxaliplatin), but only small proportion of them can be cured, usually with subsequent consolidation surgery. At that stage the disease is usually chemorefractory and there are no other chemotherapy regimens of proven benefit (7).

The purpose of this study is to determine if multiple-relapsed chemorefractory pts may benefit from sorafenib monotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. Male patients > 18 years of age
2. Patients with histologically proven germ cell neoplasm (gonadal or extragonadal primary)
3. Patients must have the disease not amendable to cure with either surgery or chemotherapy
4. Patients must have failed at least two cisplatin-based combination chemotherapy regimens.
5. Failure on prior regimens will be defined as either:

   * A ≥ 25% increase in sum of target lesions, new lesions, or
   * An increasing AFP or HCG above the nadir level.
6. Patients with at least one measurable lesion by CT scan or MRI according to RECIST criteria
7. Adequate bone marrow, liver and renal function, assessed no longer than 14 days before treatment start, defined by the following laboratory test limits: WBC > 2.0 x 109/l and platelets > 60 x 109/l, total bilirubin < 2 x upper limit, AST and ALT < 5 x upper limit normal, serum creatinine < 2 x UNL
8. WHO Performance Status 0, 1, 2
9. No concurrent chemotherapy or radiotherapy
10. Life expectancy of at least 12 weeks
11. Absence of any physiological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule
12. A signed informed consent must be obtained prior to any study specific procedures
13. All patients must agree to use adequate contraception during the whole study period

Exclusion Criteria:

1. Patients not fulfilling of inclusion criteria
2. Primary radiotherapy in the field of target lesion
3. Major surgery (RPLND) within 4 weeks before the start of study drug or concurrent serious non-healing wounds, ulcers or bone fractures.
4. Known serious and active bacterial, viral or fungal infection (> grade II CTC-AE) including HBV, HCV and HIV carrier state.
5. Previous or concurrent malignancy except for basal cell carcinoma of the skin
6. Uncontrolled hypertension.
7. Thrombotic or embolic event in last 6 months prior to inclusion.
8. Impairment of gastrointestinal tract, or GI disease that may influence the bioavailability of oral sorafenib
9. Substance and alcohol abuse (nicotine use is allowed)
10. Known or suspected hypersensitivity to sorafenib.
11. Participants in any other clinical trial using investigational drug within 4 weeks prior to study entry
12. Prior use of investigational or licensed angiogenesis and RAF kinase or MEK inhibitors.
13. Patient unwilling or unable to give informed consent
14. Any condition that may in the investigator's opinion jeopardize the safety of the patient or his compliance in the study.

Ages: 18 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2008-09; Primary Completion 2011-12 (Estimated); Study Completion 2011-12 (Estimated)

PRIMARY OUTCOMES:
Progression free survival | one year

SECONDARY OUTCOMES:
ORR Evaluation of the usefulness the CT with vasculature visualisation option in the measurement of the objective response Evaluation of quality of life | one year

CONTACTS AND LOCATIONS:
Locations (1):
- Chemotherapy Unit, Dept of Urology, Instituite of Oncology, Warsaw, Poland